CLINICAL TRIAL: NCT00655317
Title: Acupuncture and Post-Operative Ileus: A Prospective Randomized Study to Evaluate the Effects of Electrostimulated Acupuncture on Recovery From Ileus Following Standard Elective Colon Surgery
Brief Title: Acupuncture and Post-Operative Ileus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Philip P. Metzger, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 06-009410
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Ileus
Keywords: acupuncture; colon surgery; post operative ileus; post ileus; ileus; colectomy; colorectal pathology
MeSH Terms: conditions — Ileus | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Treatment Acupuncture Group (Therapeutic Acupuncture Treatment): treatment with actual acupuncture needles
  Interventions: Other: Acupuncture
- 2 (Sham Comparator): SHAM (control) acupuncture group: non-therapeutic acupuncture treatment
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Acupuncture — Treatment acupuncture group: therapeutic acupuncture treatment with actual needles
  Arms: 1
Other: Sham acupuncture — SHAM (control) acupuncture group: non-therapeutic acupuncture treatment
  Arms: 2

SUMMARY:
Postoperative ileus, the transient cessation of normal bowel function, is a universal aspect of colon surgery. Its occurrence may lead to increased patient discomfort and additional time and cost to hospital stay. Evidence from previous studies indicate that acupuncture may be beneficial in decreasing time to recovery of bowel function and decrease the body's inflammatory response. However, this has not been studied in a randomized, prospective fashion in colon surgery. The goal of this study is to determine if acupuncture may be utilized as a therapeutic modality to decrease time to return of bowel function and discharge from the hospital.

DETAILED DESCRIPTION:
The pathogenesis of post-operative ileus is not completely known. It is thought that post-operative ileus involves trauma to the bowel. This traumatizing of the intestine and peritoneal surfaces results in production and release of inflammatory mediators. These in turn, lead to inactivation of inhibitory neural reflexes. There is also an additive effect of opioids used for post-operative pain, aggravating and adding to the duration of post-operative ileus. Acupuncture has shown promise in both human and animal model studies to reduce post-operative nausea and vomiting and post-operative ileus. It is the investigator's hypothesis that acupuncture will minimize or reduce both post-operative ileus and nausea following elective colon surgery and will lead to a decrease in inflammatory markers that are known to be elevated following abdominal surgery.

The study goals are to determine if acupuncture:

* Leads to earlier return of bowel function
* Leads to earlier time to discharge following colon surgery
* Leads to earlier return of colonic motility
* Leads to decreased postoperative nausea and vomiting
* Leads to a decrease in inflammation

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age 18-89
* colorectal pathology requiring standard elective open or laparoscopic colectomy

Exclusion Criteria:

* pregnancy
* pacemaker or implantable electronic devices
* bowel obstruction
* intra-abdominal abscess or sepsis
* colorectal tumors invading other organs or surrounding tissues
* diverticulitis complicated by fistula
* known immunodeficiency disorders
* tumors requiring an anastomosis below 7cm above the anal verge as measured by rigid proctosigmoidoscope exam at surgery
* chronic pain medications
* surgeries requiring temporary or permanent ostomies
* emergent operations
* receiving preoperative radiation/chemotherapy
* major deformities of the upper or lower extremities and/or any active skin lesions or ulcers in acupunctural treatment areas

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Determine if acupuncture leads to earlier return of bowel function and earlier time to discharge following colon surgery. | Randomized acupuncture will be performed within 24 hours of completion of standard elective colon surgery

SECONDARY OUTCOMES:
Acupuncture will lead to decreased time to return of colonic motility, as measured by earlier progression of radiological markers through the colon | radiological markers will be given preoperatively and then will be tracked via abdominal x-rays postoperatively
Acupuncture will lead to decreased postoperative nausea and vomiting, resulting in less requirement of antiemetic medication | number of doses of antiemetic meds and number of episodes of vomiting and nausea will be recorded postoperatively
Acupuncture will blunt the inflammatory response, which is associated with development of postoperative ileus | serum inflammatory markers will be measured preoperatively and postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Philip P. Metzger, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota